CLINICAL TRIAL: NCT05670704
Title: A Phase 1, Randomized, Double-Blinded, Placebo-Controlled Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Immunogenicity of Single and Multiple Ascending Doses of ARGX-119 in Healthy Participants
Brief Title: A Clinical Trial to Investigate the Safety, Tolerability, Pharmacokinetics, and Immunogenicity of Single and Multiple Ascending Doses of ARGX-119 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: argenx (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: ARGX-119-2201; 2022-002529-90 (EudraCT Number)
Record Dates: First submitted 2022-12-20; First posted 2023-01-04 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ARGX-119 (Experimental): Patients receiving ARGX-119 IV or SC
  Interventions: Biological: ARGX-119
- Placebo (Placebo Comparator): Patients receiving Placebo IV or SC
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: ARGX-119 — Patients receiving ARGX-119 IV or SC
  Arms: ARGX-119
Other: Placebo — Patients receiving Placebo IV or SC
  Arms: Placebo

SUMMARY:
This phase 1 study is an FIH, double-blinded, placebo-controlled study investigating the safety, tolerability, PK, and immunogenicity of ARGX 119 administered as single doses (IV or SC) or multiple doses (IV) to healthy participants. The study IMPs are ARGX-119 or placebo for IV or SC administration.

This study will include 2 parts:

* In part A, ARGX-119 IV (or placebo IV) will be administered to 9 cohorts as single doses , while ARGX-119 SC (or placebo SC) will be administered to a 10th cohort.
* In part B, 4 once-weekly IV doses of ARGX-119 (or placebo IV) will be administered in up to 5 cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Has reached the age of consent at the time of signing the informed consent form and ≤65 years of age
* Is capable of providing signed informed consent and understands and is capable of complying with protocol requirements
* Is a healthy participant, defined as having no clinically meaningful abnormalities identified in any of the following assessments before the first IMP administration on day 1: medical history, physical examination, standard 12-lead ECG, vital sign measurements, and clinical laboratory tests
* Is either male or female of nonchildbearing potential.
* Has negative serum pregnancy tests at both screening and on day -1 (female participants)
* Has a BMI within the range of 18 to 30 kg/m2 and a body weight within the range of 50 to 100 kg (inclusive) before first IMP administration
* Agree to use contraceptive measures consistent with local regulations
* Agrees to discontinue and refrain from using all medications, including nonprescription and prescription medications, for ≥2 weeks before their first IMP administration through the study. The occasional use of paracetamol is allowed upon approval by the investigator.
* Is a nonsmoker (defined as an individual who has abstained from smoking for ≥3 months before screening) and does not use nicotine-containing products
* Has a negative drug and alcohol test for amphetamines, barbiturates, benzodiazepines, cannabis, cocaine, opiates, methadone, tricyclic antidepressants, and alcohol at screening and on day -1
* Has a body temperature of 35.5 °C to 37.6 °C at screening and before their first IMP administration on day 1

Exclusion Criteria:

* Has a known hypersensitivity to any of the components of the IMP, or has a history of a significant allergic reaction to any drug that is considered exclusionary by the investigator
* Has been given an investigational product within 3 months or 5 half-lives (whichever is longer) before their first IMP administration
* Has a positive serum test at screening for an active infection with any of the following conditions: HBV that is indicative of an acute or chronic infection, unless associated with a negative HBsAg or negative HBV DNA test, HCV based on HCV antibody assay unless a negative RNA test is available, HIV based on test results
* Has a positive COVID-19 test result on day -1, if performed.
* Has a history of any medical or psychiatric condition that, in the opinion of the investigator, is clinically meaningful, may confound the result of the study, or may pose additional risks to the participant while taking part in the study
* Has clinically relevant abnormalities detected on an ECG that are related to either rhythm or conduction
* Has a clinically meaningful abnormality in any screening test or vital sign measurement before their first IMP administration
* Has had an event causing significant blood loss (including blood donation >500 mL) or a transfusion of any blood product ≤12 weeks before their first IMP administration
* Has a history of any of the following: Consuming >21 units of alcoholic beverages per week ≤2 years before screening; Alcoholism or drug, chemical, or substance abuse ≤2 years before screening; Consuming a large quantity (>6 cups a day) of coffee, tea, or equivalent during the 4 week screening period
* Has any condition that impairs phlebotomy, including (but not limited to) coagulation disorders (hemophilia A, hemophilia B, Von Willebrand disease), clotting factor deficiencies, or any other condition that would increase the risk of hematoma formation
* Is an investigator, subinvestigator, research assistant, pharmacist, study coordinator, or other staff or relative of study personnel directly involved with the conduct of the study
* Has any condition or circumstances that, in the opinion of the investigator, may make a participant unlikely or unable to complete the study or comply with study procedures and requirements

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2023-02-21 (Actual); Primary Completion 2024-08-08 (Actual); Study Completion 2024-08-08 (Actual)

PRIMARY OUTCOMES:
Number of treatment-emergent adverse events (TEAEs) | up to 157 days for part A, 117 days for part B

SECONDARY OUTCOMES:
Pharmacokinetic parameters of ARGX-119: Area Under The Curve (AUC) | up to 157 days for part A, 117 days for part B
Pharmacokinetic parameters of ARGX-119: Maximum serum concentrations (Cmax) | up to 157 days for part A, 117 days for part B
Pharmacokinetic parameters of ARGX-119: Time to reach maximum serum concentrations (Tmax) | up to 157 days for part A, 117 days for part B
Incidence of antidrug antibodies against ARGX-119 | up to 157 days for part A, 117 days for part B

CONTACTS AND LOCATIONS:
Locations (1):
- PRA Health Science, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided